CLINICAL TRIAL: NCT04039711
Title: Evaluation of Vaginal Self-sampling Diagnostic Performances to Identify Genital Infections : A Large, Cross-sectional, Non-inferiority Trial
Brief Title: Evaluation of Vaginal Self-sampling Diagnostic Performances to Identify Genital Infections
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hôpital Européen Marseille (Other)
Responsible Party: Principal Investigator, Edwin QUARELLO @me.com, Principal investigator, Hôpital Européen Marseille
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RCB 2014-A01250-47
Record Dates: First submitted 2019-07-29; First posted 2019-07-31 (Actual); Last update posted 2019-08-02 (Actual); Status verified 2019-08

CONDITIONS: Genital Infection; Asymptomatic Infections
Keywords: Vaginal self-sampling; STI; Genital infection; Group B streptococcus
MeSH Terms: conditions — Asymptomatic Infections; Sexually Transmitted Diseases

STUDY DESIGN:
Intervention Model Description: Participants were screenned for genital infections
  * performing vaginal and/or cervical classical-sampling (VCS)
  * performing vaginal self-sampling (VSS)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Genital infections (Other): Women with vaginal/cervical sampling indications
  Interventions: Procedure: Vaginal self-sampling

INTERVENTIONS:
Procedure: Vaginal self-sampling — The objective is to determine the non-inferiority of vaginal self-sampling compared with vaginal/cervical classical sampling, and evaluate the possibility of using it in all clinical situations indicating the prescription of such a procedure to screen for genital infections (GIs), sexually transmitted infections (STIs) and group B streptococcus (GBS) asymptomatic carriage in pregnant women.

SUMMARY:
Screening for genital infection (GI), sexually transmitted infection (STI) and asymptomatic carriage of group B streptococcus (GBS) in pregnant women is a common reason for medical appointments. Conventional testing is performed by using vaginal and/or cervical classic sampling (VCS). Vaginal self-sampling (VSS) has progressively emerged as an alternative to VCS for STI agent screening. The use of vaginal self-sampling (VSS) could facilitate follow-ups and potentially help in the prevention of gynaecological disorders.

ELIGIBILITY:
Inclusion Criteria:

* Women requiring vaginal or cervical classical sampling to screen for genital infections
* Women requiring vaginal or cervical classical sampling to screen for sexually transmitted infections (STI)
* Pregnant women requiring vaginal classical sampling to screeen for Group B streptococcus asymptomatic carriage in the eighth month of pregnancy
* Informed written consent from the patient

Exclusion Criteria:

* Person subjected to therapeutic limitation decision
* Women with intact hymen
* Active antibiotic or antifungic treatment
* Antiobiotic or antifungic treatment during the 10 days prior to inclusion

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 1028 (Actual)
Dates: Start 2015-10-20 (Actual); Primary Completion 2018-04-06 (Actual); Study Completion 2018-04-06 (Actual)

PRIMARY OUTCOMES:
Bacterial infection detection rates | 10 days
  Bacterial infection detection rates of VSS compared with VCS
Yeast infection detection rates | 10 days
  Yeast infection detection rates of VSS compared with VCS
Chlamydia trachomatis detection rates | 10 days
  Chlamydia trachomatis detection rates of VSS compared with VCS
Neisseria gonorrhoeae detection rates | 10 days
  Neisseria gonorrhoeae detection rates of VSS compared with VCS
Mycoplasma genitalium detection rates | 10 days
  Mycoplasma genitalium detection rates of VSS compared with VCS
Trichomonas vaginalis detection rates | 10 days
  Trichomonas vaginalis detection rates of VSS compared with VCS
Human simplex virus detection rates | 10 days
  Human simplex virus detection rates of VSS compared with VCS
Group B streptococcus detection rates | 10 days
  Group B streptococcus detection rates of VSS compared with VCS

CONTACTS AND LOCATIONS:
Locations (1):
- European Hospital, Marseille, Bouches-du Rhone, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hobbs MM, van der Pol B, Totten P, Gaydos CA, Wald A, Warren T, Winer RL, Cook RL, Deal CD, Rogers ME, Schachter J, Holmes KK, Martin DH. From the NIH: proceedings of a workshop on the importance of self-obtained vaginal specimens for detection of sexually transmitted infections. Sex Transm Dis. 2008 Jan;35(1):8-13. doi: 10.1097/OLQ.0b013e31815d968d. PMID 18157061
- [Result] Lunny C, Taylor D, Hoang L, Wong T, Gilbert M, Lester R, Krajden M, Ogilvie G. Self-Collected versus Clinician-Collected Sampling for Chlamydia and Gonorrhea Screening: A Systemic Review and Meta-Analysis. PLoS One. 2015 Jul 13;10(7):e0132776. doi: 10.1371/journal.pone.0132776. eCollection 2015. PMID 26168051